CLINICAL TRIAL: NCT02214264
Title: Brief Trainings to Buffer Against Acute Stress Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-0572; MLK2014 (Other: Study Team)
Record Dates: First submitted 2014-07-31; First posted 2014-08-12 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Loving-Kindness training (Experimental): Participants receive Loving-Kindness meditation training for approximately 12 minutes.
  Interventions: Behavioral: Loving-Kindness meditation training
- Breath Awareness training (Experimental): Participants receive Breath Awareness meditation training for approximately 12 minutes.
  Interventions: Behavioral: Breath Awareness meditation training
- Gratitude training (Experimental): Participants will receive Gratitude training for approximately 12 minutes.
  Interventions: Behavioral: Gratitude
- Control (Other): Participants write and then think about the physical space in which they live (i.e., their home) for approximately 12 minutes.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Loving-Kindness meditation training — Participants undergo training for approximately 12 minutes. Training involves guided reflections and intentions related to feeling loving-kindness towards the self and others.
  Arms: Loving-Kindness training
Behavioral: Breath Awareness meditation training — Participants undergo training for approximately 12 minutes. Training involves guided awareness focused on sensations of breathing.
  Arms: Breath Awareness training
Behavioral: Gratitude — Participants undergo training for approximately 12 minutes. Training involves reflections of gratitude for people, events, and things in one's life.
  Arms: Gratitude training
Behavioral: Control — Participants will write and then think about the physical space in which they live (i.e., their home) for approximately 12 minutes.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate and compare the effectiveness of several brief trainings based on contemplative practices and positive psychology to buffer against the negative effects that acute stress has on behavior and cognitive abilities. The investigators hypothesize that training will buffer against negative effects of acute stress.

DETAILED DESCRIPTION:
Participants will be taught a stress reducing training (breath awareness, loving kindness practice, gratitude exercise) and will practice using this technique for 10-15 minutes. Following this, all participants will undergo the Cold Pressor Task (CPT) for up to 3 minutes.

Before and after these tasks, participant data related to attention, working memory, self regulation, affect, and prosociality will be collected.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate psychology recruitment pool

Exclusion Criteria:

* non-native English speakers, pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline performance on Operational Span task | Baseline and 10 minutes following post stress induction
Change from baseline in time spent on hand grip self regulation task | Baseline and 30 minutes post stress induction
Change from baseline on likeability ratings of neutral stimuli | Baseline and 1 minute post stress induction
Number of trials completed in optional Generosity task | 40 minutes post stress induction
Positive and Negative Affect Schedule ratings at baseline | Baseline
Positive and Negative Affect Schedule ratings after pre-test measures | 2 minutes before training
Positive and Negative Affect Schedule ratings after training | 1 minute after training
Positive and Negative Affect Schedule ratings after stress induction | 1 minute after stress induction
Positive and Negative Affect Schedule ratings after post-test | 1 minute after post-test measures
Implicit Positive and Negative Affect Test at baseline | Baseline
Implicit Positive and Negative Affect Test after pre-test measures | 2 minutes before training
Implicit Positive and Negative Affect Test after training | 1 minute after training
Implicit Positive and Negative Affect Test after stress induction | 1 minute after stress induction
Implicit Positive and Negative Affect Test after post-test | 1 minute after post-test

SECONDARY OUTCOMES:
Participant interest in participating in future training | 40 minutes post stress induction
  Interest will be rated using a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Schaefer, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Goldberg SB, Flook L, Hirshberg MJ, Davidson RJ, Schaefer SM. Brief breath awareness training yields poorer working memory performance in the context of acute stress. Cogn Emot. 2021 Aug;35(5):1009-1017. doi: 10.1080/02699931.2021.1878113. Epub 2021 Jan 29. PMID 33509056